CLINICAL TRIAL: NCT03434496
Title: The Role of Music in Improving Gait Abnormalities in Parkinson Disease
Brief Title: Music Role in PD Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, MD PhD, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/2017
Record Dates: First submitted 2018-01-31; First posted 2018-02-15 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-02

CONDITIONS: Parkinson Disease
Keywords: PD; Gait training 3; treadmill.
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental group (Experimental): The investigators will enroll 30 patients with PD, randomly divided into two groups: (A) gait training with Music; (B) conventional treadmill gait training. The 15 patients in the experimental group will perform training by means of the device Gait Trainer 3 (Biodex), where they will train on a tredmill equipped with music. They will walk following specific musical beets and rhythms so to entrain their own internal rhythm. Subjects will attend 3 sessions a week for at least 4 weeks. Each session will last 45-min.
  Interventions: Device: Gait Trainer 3
- Control Group (Active Comparator): The control group will perform only conventional gait treadmill training, besides physical exercises to improve muscle force and tone. Subjects will attend 3 sessions a week for at least 4 weeks. Each session will last 45-min.
  Interventions: Device: Gait Trainer 3

INTERVENTIONS:
Device: Gait Trainer 3 — With the BIODEX Gait Trainer 3, patients acquire a smooth gait pattern. In addition, balance, coordination, endurance and the cardiovascular system are trained. Work on the treadmill strengthens the leg muscles. On the screen or via an audio message, the patients and therapists receive direct feedback on the smoothness of the gait pattern. The therapists can then make corrective interventions if necessary and the patients are motivated.
  Other Names: Conventional physioterapy

SUMMARY:
Neurologic Music Therapy (NMT) sensorimotor techniques are increasingly used to improve spatio-temporal gait parameters and postural stability in the course of Parkinson's Disease and following stroke. Nonetheless, the neurophysiological underpinnings of NMT-mediated gait recovery is still poorly understood.

The aim of the study was to investigate the central mechanisms of connectivity related to the application of Rhythmic Auditory Stimulation (RAS) in PD gait rehabilitation. The investigators will enroll 30 patients with PD. They will be randomized into two groups: (A) gait training with Music; (B) conventional treadmill gait training. The experimental group will perform training by means of GT3 (Biodex), where the patient is able to walk (on a treadmill) following specific musical beets and rhythms. The control group will perform only gait treadmill training.

Subjects will attend 3 sessions a week for at least 4 weeks. Each session will last 45-min.

DETAILED DESCRIPTION:
The aim of the study was to investigate the central mechanisms of connectivity related to the application of Rhythmic Auditory Stimulation (RAS) in PD gait rehabilitation. The investigators will enroll 30 patients with PD. They will be randomized into two groups: (A) gait training with Music; (B) conventional treadmill gait training. The experimental group will perform training by means of GT3 (Biodex), where the patient is able to walk (on a treadmill) following specific musical beets and rhythms. The control group will perform only gait treadmill training.

Subjects will attend 3 sessions a week for at least 4 weeks. Each session will last 45-min.

The investigators will assess the gait performance and pattern by using System BTS Smart for gait and the sensorimotor functional connectivity by using EEG, both before and after the therapy cycle. The patients will be clinically evaluated by means of Time up and go test, and ten meters. The overall motor function will be evaluated through the UPDRS III.

Power calculation by Cohen (1992) methodology will be utilized for this pilot study. Shapiro-Wilk test was applied to assess the normality of distribution. Thus, parametric and non-parametric tests will be employed for all comparisons (Wilcoxon test, ANOVA). Mann-Whitney test or ANOVA will be utilized to evaluate the level of significance in differentiation between the examined groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by PD;
* MMSE > 21
* Hoehn and Yahr <3

Exclusion Criteria:

* Presence of severe cognitive deficit
* Severe motor impairment (Hoehn and Yahr >3)
* Medical illness potentially interfering with the training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Ten meters walking test | about 4 weeks
  It is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.

SECONDARY OUTCOMES:
Electroencephalogram | about 4 weeks
  It can be employed to evaluate the improvement in functional connectivity, i.e. the dinamic relation between different brain areas.

CONTACTS AND LOCATIONS:
Overall Officials: Placido Bramanti, MD, Study Director — IRCCS Neurolesi
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calabro RS, Naro A, Filoni S, Pullia M, Billeri L, Tomasello P, Portaro S, Di Lorenzo G, Tomaino C, Bramanti P. Walking to your right music: a randomized controlled trial on the novel use of treadmill plus music in Parkinson's disease. J Neuroeng Rehabil. 2019 Jun 7;16(1):68. doi: 10.1186/s12984-019-0533-9. PMID 31174570